CLINICAL TRIAL: NCT04362514
Title: "Safer Cycling in Older Age" - a Multi-component Exercise Intervention in Community-dwelling, Older Adults.
Brief Title: Safer Cycling in Older Age
Acronym: SiFAr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: ADAC (The General German Automobile Club) foundation (Unknown)
Responsible Party: Principal Investigator, Robert Kob, PhD, Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBA-2020-SiFAr
Record Dates: First submitted 2020-04-14; First posted 2020-04-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2022-12

CONDITIONS: Older Adults; Community-dwelling; Cycling Competence
Keywords: Older cyclists; Bicycling; Multi-component exercise; Motor competence; Stress; Psychological concerns

STUDY DESIGN:
Intervention Model Description: SiFAr is a parallel group, randomized controlled trial with a duration of 3 years and a recruitment period between June 2020 and July 2022. The 1:1 randomization of participants to IG or aCG is stratified by gender and bicycle type (e-bikes/unmotorized bicycle).
  Baseline data collection (T0) takes place in-person in the study center and in the cycle course on two different days within approximately 14 days. Except for cognitive function, same data are collected of all participants after the 3 months intervention period (T1), regardless of their compliance. In addition, participants will be followed up 6-9 months after T1 (T2) related to seasonal time frames (after winter season). Furthermore, participants of the IG 2020 will be measured for a long-term follow-up in the third year of the study (T3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IG (Experimental): Intervention Group
  Interventions: Behavioral: MEPC - Multi-component exercise program related to cycling
- aCG (Active Comparator): Control Group
  Interventions: Other: HRP - health-related presentations

INTERVENTIONS:
Behavioral: MEPC - Multi-component exercise program related to cycling — Structured and progressive multicomponent exercise program with and without bikes. Training period will last over 3 months with 8 sessions à 60 minutes. Training sessions will address motor competence (balance, strength, cycling skills and techniques) and cognitive skills required during cycling. Furthermore, fall-related psychological concerns will be addressed.
  Arms: IG
Other: HRP - health-related presentations — HRP include 3 presentations on healthy aging (one per month) with a duration of 60 minutes
  Arms: aCG

SUMMARY:
The aim of the SiFAr-project is to increase safe cycling in community-dwelling older adults (age 65 years and older) with a structured, multi-component exercise cycling training. The progressive exercise program encompasses training of motor competence and cognitive functions. The ability to cycle safely will be tested prior and after the training period using a cycling course, which consists of variant tasks requiring motor and cognitive skills.

DETAILED DESCRIPTION:
Cycling is a form of physical activity that is positively associated with health and functional benefits. In Germany, the use of bicycles, especially of those with motorized assistance (e-bikes), is steadily increasing among older adults. Despite the benefits mentioned, cycling also poses potential health risks. For instance, there is a significant association between increased bicycle use and bicycle crashes. This relationship is particularly evident in older adults with a higher prevalence of bicycle crashes leading to minor and serious injuries. This might be explained by the age-related decline of physical and cognitive function, which may essentially affect (reduce) the ability to cycle safely. In order to prevent crashes and falls from bicycles, targeted training of the required skills for safe cycling could be effective. However, there is a lack of scientifically evaluated bicycle-training concepts that have been developed specifically for older adults.

By developing and providing a structured and progressive multi-component exercise program related to cycling for older adults, the SiFAr-project will address the improvement of bicycle-related basic motor competence (e.g. balance, strength, ability to react, cycling skills and techniques) and the reduction of stress and fall-related psychological concerns.

The ability to ride a bike safely will be measured in both arms before and after the training period by completing various tasks in a cycling course.

The aim of the program is that the participation in the three-month exercise intervention program will lead to a reduction of failures in the bicycle course. As comparative values, the number of faults in the bicycle course before the training period and the number of faults in the control group will be used. Furthermore, a substudy aim to investigate stress biomarkers targeting inflammatory and stress associated physiological parameters during cycling. The activity of stress systems will be determined by measuring stress hormones like cortisol and inflammatory responses in the body by measuring C-reactive protein. To analyse biomarkers, saliva, hair and blood specimen will be collected.

ELIGIBILITY:
Inclusion Criteria:

* living in the area Nürnberg-Fürth-Erlangen, Bavaria, Germany
* Ability to come to training locations on their own bicycle, having a suitable helmet
* participant is either 1) a beginner with the e-bike or has 2) self-reported insecurity or is 3) a re-entrant in cycling

Exclusion Criteria:

* long-term, experienced cyclists without subjectively reported limitations or worries when cycling.
* diseases that contradict safe participation in the intervention (e.g. myocardial infarction within the last 6 months, unstable angina pectoris, cerebrovascular event, serious cancer diagnosis, serious neurological diseases like Parkinson, dementia; and other serious new diagnosis)
* other factor that prevent regular and safe participation in the intervention (e.g. prolonged holidays during the training period, alcoholism)
* severe visual impairments that cannot be sufficiently compensated by a visual aid

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Number of faults in the cycling course | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  The cycling competence will be tested in a standardized cycling course, including the following tasks: slalom, slow cycling within a marked lane, dismounting into a marked zone, getting on the bike, cycling through a narrow alley, turning to the off-side, braking with pinpoint accuracy. Mean change of number of faults in the cycling course will be tested between pre- and postintervention.

OTHER OUTCOMES:
Short Physical Performance Battery (SPPB) | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  mean change in sumscore (0-12 points)
Fear of Falling (Short FES-I) | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  mean change in sumscore (7-28 points)
Cortisol | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  change in concentration in nmol/L by high-sensitive Enzyme-linked Immunosorbent Assay (ELISA)
Alpha-amylase | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  change in concentration in enzyme units U/mL by Enzyme kinetic Assay
C-reactive protein (CRP) | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  change in concentration in mg/L by high-sensitive Enzyme-linked Immunosorbent Assay (ELISA)
EuroQol (EQ-5D) | changes over a period of 3 months and after a follow-up period of 6-9 and in some cases 18-21 months
  change in sumscore and change in mean value of Visual-Analogue-Scale (VAS, 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kob, PhD, Principal Investigator — Institute for Biomedicine of Aging
Locations (1):
- Institute for Biomedicine of Aging, Nuremberg, Bavaria, Germany

REFERENCES:
- [Background] Siebentritt HM, Keppner V, Britting S, Kob R, Rappl A, Sieber CC, Freiberger E. Safer cycling in older age (SiFAr): a protocol of a randomized controlled trial. BMC Geriatr. 2021 Oct 12;21(1):546. doi: 10.1186/s12877-021-02502-5. PMID 34641821
- [Background] Keppner V, Krumpoch S, Kob R, Rappl A, Sieber CC, Freiberger E, Siebentritt HM. Safer cycling in older age (SiFAr): effects of a multi-component cycle training. a randomized controlled trial. BMC Geriatr. 2023 Mar 7;23(1):131. doi: 10.1186/s12877-023-03816-2. PMID 36882759
- [Background] Keppner V, Sieber CC, Freiberger E, Kob R, Krumpoch S, Siebentritt HM. Characteristics of older cyclists with self-perceived needs for improvement in cycling competence: SiFAr trial. Eur Geriatr Med. 2023 Jun;14(3):595-602. doi: 10.1007/s41999-023-00765-2. Epub 2023 Mar 28. PMID 36973532
- [Derived] Britting S, Kob R, Sieber CC, Rohleder N, Freiberger E, Becker L. Physiological stress in safer cycling in older age (SiFAr-stress): effect of a multicomponent exercise intervention-a study protocol for a randomized controlled trial. Trials. 2021 Aug 21;22(1):552. doi: 10.1186/s13063-021-05481-5. PMID 34419134